CLINICAL TRIAL: NCT04525352
Title: A Phase I Clinical Trial for Gene Therapy in Infantile Malignant Osteopetrosis (IMO) to Evaluate the Safety and Preliminary Efficacy of Autologous CD34+ Enriched Cells Transduced With a LV Vector Encoding the TCIRG1 Gene
Brief Title: A Trial to Evaluate Safety and Efficacy of RP-L401-0120 in Subjects With Infantile Malignant Osteopetrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study discontinued due to feasibility.
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-L401-0120
Record Dates: First submitted 2020-08-11; First posted 2020-08-25 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Infantile Malignant Osteopetrosis
Keywords: Impaired bone resorption; Deficient osteoclast development; Autosomal Recessive Disorder; Musculoskeletal Diseases; Bone Diseases; Hypocalcemia; Bone marrow failure
MeSH Terms: conditions — Musculoskeletal Diseases; Bone Diseases; Hypocalcemia; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental - RP-L401 (Experimental): RP-L401 is a gene therapy product containing autologous genetically modified CD34+ hematopoietic cells transduced with lentiviral vector carrying the TCIRG1 transgene
  Interventions: Biological: RP-L401

INTERVENTIONS:
Biological: RP-L401 — CD34+ enriched hematopoietic stem cells from pediatric subjects with infantile malignant osteopetrosis transduced ex vivo with lentiviral vector carrying the TCIRG1 transgene

SUMMARY:
The primary objective of this Phase 1 study is to evaluate the therapeutic safety and feasibility of the investigational product (IP), RP-L401.

DETAILED DESCRIPTION:
This is a non-randomized Phase 1 study to evaluate the preliminary safety and efficacy of hematopoietic gene therapy consisting of autologous CD34+ enriched hematopoietic cells transduced with the lentiviral vector (LV) carrying the human TCIRG1 transgene (RP-L401) in pediatric patients with IMO. Following myeloablative conditioning patients will receive an infusion of the genetically modified hematopoietic stem and progenitor cells (HSPCs).

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of IMO with documented TCIRG1 mutation.
2. Age at least 1 month with minimum weight of 4 kg
3. Absence of debilitating hydrocephalus (defined as hydrocephalus at NCI CTCAE v5.0 Grade 3 or higher persisting despite shunt or similar procedural intervention).
4. Lansky Play Scale of at least 60%
5. Preserved hepatic function (AST/ALT ≤3.0 ULN; bilirubin ≤1.5 ULN; to minimize potential for excessive toxicity from busulfan conditioning)
6. No concomitant medical or other conditions that would represent a contraindication to autologous hematopoietic stem cell transplant.
7. Absolute neutrophil count of ≥500/mm3 and platelet count of ≥25,000/mm3
8. No prior allogeneic or other hematopoietic stem cell transplant.
9. Availability of a non-autologous rescue (back-up) hematopoietic stem cell donor/source

Exclusion Criteria:

1. Availability of medically-feasible HLA-matched sibling donor for allogeneic HSCT.
2. Any medical or other contraindication for either apheresis or autologous transplant as determined by the Investigator.
3. Participation in another clinical trial with an investigational drug within 14 days before the informed consent signature. Participation in observational studies is allowed.
4. Active hematologic or solid organ malignancy, not including non-melanoma skin cancer or another carcinoma in situ.
5. Uncontrolled seizure disorder.
6. Renal dysfunction as defined by a glomerular filtration rate <30 mL/min/1.73m2 or dialysis dependence.
7. Serious infections with persistent bloodstream pathogens at time of trial entry
8. Pulmonary dysfunction as defined by either:

   * Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection) or
   * Oxygen saturation (by pulse oximetry) <90% resulting from pulmonary conditions (intermittent hypoxia secondary to IMO-related choanal atresia will not be considered exclusionary)

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 2 years
  Evaluation of safety associated with treatment with RP-L401

SECONDARY OUTCOMES:
Assessment of vector copy number (VCN) after infusion of RP-L401 | 2 years
  Evaluation of the presence of gene-modified blood and bone marrow cells post infusion via blood and bone marrow assessments
Assessment of endocrine and metabolic status after infusion of RP-L401 | 2 years
  Evaluation of normalization of serum calcium levels via a blood assessment
Assessment of blood counts after infusion of RP-L401 | 2 years
  Evaluation of the stabilization or improvement in blood counts as assessed by NCI CTACE
Assessment of bone abnormalities after infusion of RP-L401 | 2 years
  Evaluation of the qualitative improvement in bone formation via x-ray studies
Assessment of auditory status after infusion of RP-L401 | 2 years
  Evaluation of the stabilization or improvement in hearing loss via auditory tests
Assessment of ophthalmology status after infusion of RP-L401 | 2 years
  Evaluation of optical abnormalities via visual assessments of the eye
Assessment of hepatosplenomegaly after infusion of RP-L401 | 2 years
  Evaluation of hepatosplenomegaly improvement via abdominal ultrasound
Assessment of head, mouth and gum abnormalities | 2 years
  Photographic documentation of head, mouth and gums to assess disease stabilization, progression or improvement

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Kohn, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States